CLINICAL TRIAL: NCT03083548
Title: The Nor-Hand Study: An Observational Cohort of Hand Osteoarthritis Patients
Brief Title: The Nor-Hand Study
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Ida Kristin Haugen, MD, PhD, Diakonhjemmet Hospital
Other Study IDs: DIA2017-1
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Pain; Inflammation; Image, Body
MeSH Terms: conditions — Osteoarthritis; Pain; Inflammation | interventions — Diagnostic Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, urine, plasma and whole-blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hand osteoarthritis: Men and women (40-70 years) with a diagnosis of hand OA based on clinical or ultrasound examination are included. Patients with systemic inflammatory joint diseases, psoriasis and hemochromatosis are excluded.
  Interventions: Diagnostic Test: Imaging; Diagnostic Test: Physical examinations; Diagnostic Test: Questionnnaires

INTERVENTIONS:
Diagnostic Test: Imaging — Conventional radiographs (hands/feet), CT of dominant hand, MRI of dominant hand, ultrasound (hands/shoulder/feet/hips/knees), fluorescence optical imaging of hands
Diagnostic Test: Physical examinations — Joint assessment of hands and feet, pain sensitization test and functional tests
Diagnostic Test: Questionnnaires — Self-reported demographic factors, clinical variables and OA history and symptoms

SUMMARY:
The Nor-Hand study is a hospital-based observational study including 300 patients with evidence of hand OA by ultrasound and/or clinical examination. The baseline examination (2016-17) consists of functional tests and joint assessment of the hands, medical assessment, pain sensitization tests, ultrasound (hands, acromioclavicular joint, hips, knees and feet), computer tomography (CT) and Magnetic Resonance Imaging (MRI) of the dominant hand, conventional radiographs of the hands and feet, fluorescence optical imaging of the hands, collection of blood and urine samples as well as self-reported demographic factors and OA-related questionnaires. Two follow-up examinations are planned after 3 (2019-20) and 8 years (2024-25), respectively. Cross-sectional analyses will be used to investigate agreements and associations between different relevant measures at the baseline examination, whereas the longitudinal data will be used for evaluation of predictors for clinical outcomes and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-70 years at screening
* Proven hand OA by clinical examination and/or ultrasound

  1. Clinical examination criteria: Heberden/Bouchards nodes and/or bony enlargement, squaring and/or deformity of the thumb base and no clinical signs of inflammatory arthritis (e.g. soft tissue swelling of two or less metacarpophalangeal (MCP) joints, and no soft tissue swelling of the wrist).
  2. Ultrasound criteria: Osteophytes in the interphalangeal joints and/or the thumb base, and no signs of inflammatory arthritis (e.g. synovitis with power Doppler activity in two or less MCP joints and no synovitis with power Doppler activity in the wrist).
* Capable of understanding and signing an informed consent form
* Provided a written informed consent to participate in the study

Exclusion Criteria:

* Diagnosis of inflammatory arthritic disease, e.g. seropositive or seronegative rheumatoid arthritis, psoriatic arthritis, reactive arthritis, spondyloarthritis or arthritis related to connective tissue disorders
* Diagnosis of psoriasis
* Erythrocyte sedimentation rate (ESR) > 40 mm/hour and/or C-reactive protein (CRP) >20 mg/L, without a known ongoing infection
* Anti Cyclic Citrullinated Protein (anti-CCP) and/or rheumatoid factor positivity
* Ferritin >200 microgram/L for women and >300 microgram/L for men and s-iron/s-total iron binding capacity (TIBC) above 50%
* Major co-morbidities (e.g. severe malignancies, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease or severe respiratory disease)
* Mental or psychiatric disorders, alcohol or drug abuse, language difficulties or other factors that make compliance to the study protocol difficult.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and women between the ages of 40-70 years. Their diagnosis of hand OA has been proven either by ultrasound and/or clinical examination performed by a rheumatologist at the Rheumatology Outpatient clinic at Diakonhjemmet Hospital. In addition, all patients must be able to sign and understand an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Demographic factors | Baseline
  Self-reported relationship status, education, employment, hand tasks in work/previous work, birth place
Demographic factors | 3 year follow-up
  Self-reported relationship status, social network, education, employment
Life style factors | Baseline
  Self-reported physical activity, smoking, use of alcohol (AUDIT-C)
Life style factors | 3 year follow-up
  Self-reported physical activity, smoking, use of alcohol (AUDIT-C)
Clinical disease variables | Baseline
  Self-reported year diagnosed with OA, number of years with OA symptoms, OA in family, previous injuries of hand/foot, use of medications, previous steroid injections, use of hand orthoses, use of customized tools, previous surgeries, use of alternative therapies, use of supplements, use of nature cures, use of self-help techniques
Clinical disease variables | 3 year follow-up
  Previous injuries of hand/foot, use of medications, previous steroid injections, use of hand orthoses, use of customized tools, previous surgeries, use of alternative therapies, use of supplements, use of nature cures, use of self-help techniques
EuroQol 5 dimensions | Baseline
  Self-reported mobility, self-care, usual activity, pain/discomfort, anxiety/depression
EuroQol 5 dimensions | 3 year follow-up
  Self-reported mobility, self-care, usual activity, pain/discomfort, anxiety/depression
Sleep disturbances | Baseline
  Self-reported sleep disturbances
Sleep disturbances | 3 year follow-up
  Self-reported sleep disturbances
Michigan Hand Outcomes Questionnaire (MHOQ) | Baseline
  Aesthetic damage subscale
Michigan Hand Outcomes Questionnaire (MHOQ) | 3 year follow-up
  All subscales
Localization of joint pain (homonculus) | Baseline
  Self-reported pain during the last 24 hours and previous 6 weeks
Localization of joint pain (homonculus) | 3 year follow-up
  Self-reported pain during the last 24 hours and previous 6 weeks
Self-reported joint pain, hand pain, feet pain, fatigue, disease activity | Baseline
  Numeric Rating Scale (0-10)
Self-reported joint pain, hand pain, feet pain, fatigue, disease activity | 3 year follow-up
  Numeric Rating Scale (0-10)
Australian/Canadian hand index (AUSCAN) | Baseline
  Self-reported hand pain, stiffness and physical function
Australian/Canadian hand index (AUSCAN) | 3 year follow-up
  Self-reported hand pain, stiffness and physical function
Western Ontario and McMaster Universities Arthrtis Index (WOMAC) | Baseline
  Self-reported knee/hip pain, stiffness and physical function
Western Ontario and McMaster Universities Arthrtis Index (WOMAC) | 3 year follow-up
  Self-reported knee/hip pain, stiffness and physical function
Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) | Baseline
  Modified version to assess constant and intermittent pain in patients with hand OA (self-reported)
McGill Questionnaire | Baseline
  Modified version to assess hand OA pain characteristics (self-reported)
PainDetect | Baseline
  Modified version to assess neuropathic hand pain (self-reported)
PainDetect | 3 year follow-up
  Modified version to assess neuropathic hand pain (self-reported)
Brief Approach/Avoidance Coping Questionnaire (BACQ) | Baseline
  Self-reported approach-oriented and avoidance oriented coping
Pain catastrophizing scale | Baseline
  Self-reported magnification, rumination, helplessness
Pain catastrophizing scale | 3 year follow-up
  Self-reported magnification, rumination, helplessness
Self-efficacy scales | Baseline
  Self-reported ability influence pain and symptoms
Self-efficacy scales | 3 year follow-up
  Self-reported ability influence pain and symptoms
Foot Function Index | Baseline
  Self-reported pain in feet, disability, activity restrictions
Foot Function Index | 3 year follow-up
  Self-reported pain in feet, disability, activity restrictions
Hormonal factors in women | Baseline
  Menopause
Hormonal factors in women | 3 year follow-up
  Menarche, menopause, gynecological operations, hormone treatment, pregnancies, breastfeeding
Use of shoewear | 3 year follow-up
  The use of shoes with varying type of forefoot and heels
Global health assessment | 3 year follow-up
  The evaluation of the global health on Visual analogue scale (VAS)
Pain Sensitivity Questionnaire | 3 year follow-up
  Pain in different daily-life situations, normally leading to no or little pain
Fibromyalgia symptoms | 3 year follow-up
  ACR criteria for fibromyalgia
Short form 12 Energy | 3 year follow-up
  One question from Short form 12 about poor energy
Brief Illness Perception Questionnaire | 3 year follow-up
  Illness perception related to their hand OA disease and symptoms
Height | Baseline
  Examination of height in standing position (performed by medical student)
Height | 3 year follow-up
  Examination of height in standing position (performed by medical student)
Weight | Baseline
  Examination of weight in light-weighted clothes (performed by medical student)
Weight | 3 year follow-up
  Examination of weight in light-weighted clothes (performed by medical student)
Hip/waist circumference | Baseline
  Examination of hip and waist circumference (performed by medical student)
Hip/waist circumference | 3 year follow-up
  Examination of hip and waist circumference (performed by medical student)
Blood pressure | Baseline
  Examination of blood pressure after rest (performed by medical student)
Blood pressure | 3 year follow-up
  Examination of blood pressure after rest (performed by medical student)
Heart rate | Baseline
  Examination heart rate after rest (performed by medical student)
Heart rate | 3 year follow-up
  Examination heart rate after rest (performed by medical student)
Comorbidity questionnaires and medications | Baseline
  Self-reported comorbidities and medications
Comorbidity questionnaires and medications | 3 year follow-up
  Self-reported comorbidities and medications
Hair sample | Baseline
  Small hair sample is collected from the back of the patients´ head for quantification of cortisol
Joint assessment (examination by rheumatologist) | Baseline
  Bony enlargement, tenderness (Doyle index in hand) and soft tissue swelling in hands and feet, and assessment of the ACR criteria of hand, knee and hip
Joint assessment (examination by rheumatologist) | 3 year follow-up
  Bony enlargement, tenderness (Doyle index in hand) and soft tissue swelling in hands and feet, and assessment of the ACR criteria of hand, knee and hip
Grip strength | Baseline, follow-up
  Bilateral measurement of grip strength using Jamar dynamometer
Grip strength | 3 year follow-up
  Bilateral measurement of grip strength using Jamar dynamometer
Moberg Pick-Up test | Baseline
  Bilateral measurement of fine motor acitivities (time to pick up small elements and put in the box)
Moberg Pick-Up test | 3 year follow-up
  Bilateral measurement of fine motor acitivities (time to pick up small elements and put in the box)
Chair Stand test | 3 year follow-up
  Number of chair stands during 30 sec
40 m walking test | 3 year follow-up
  Time in sec for 40 m walking
Pain sensitization tests | Baseline
  Temporal summation, pressure pain threshold (painful finger joint, non-painful finger joint, trapezius muscle, left distal radioulnar joint and tibialis anterior muscle), conditioned pain modulation, light touch
Pain sensitization tests | 3 year follow-up
  Temporal summation, pressure pain threshold (painful finger joint, non-painful finger joint, trapezius muscle, left distal radioulnar joint and tibialis anterior muscle), conditioned pain modulation, light touch
Ultrasound examination | Baseline
  Osteophytes, grey-scale synovitis and power doppler activity in hands, AC joint, hips, knees and feet
Ultrasound examination | 3 year follow-up
  Osteophytes, grey-scale synovitis and power doppler activity in hands, AC joint, hips, knees and feet
Fluorescence Optical Imaging | Baseline
  Examination of altered microcirculation in the hands
Fluorescence Optical Imaging | 3 year follow-up
  Examination of altered microcirculation in the hands
Conventional radiographs | Baseline
  Hands (frontal), feet (frontal, oblique and side images)
Conventional radiographs | 3 year follow-up
  Hands (frontal), feet (frontal, oblique and side images)
MRI | Baseline
  MRI of dominant hand
MRI | 3 year follow-up
  MRI of dominant hand
CT | Baseline
  CT of dominant hand
Biobank | Baseline
  Collection of whole blood, serum, plasma and urine
Biobank | 3 year follow-up
  Collection of whole blood, serum, plasma and urine

CONTACTS AND LOCATIONS:
Overall Officials: Ida K Haugen, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fjellstad CM, Mathiessen A, Slatkowsky-Christensen B, Kvien TK, Hammer HB, Haugen IK. Associations Between Ultrasound-Detected Synovitis, Pain, and Function in Interphalangeal and Thumb Base Osteoarthritis: Data From the Nor-Hand Cohort. Arthritis Care Res (Hoboken). 2020 Nov;72(11):1530-1535. doi: 10.1002/acr.24047. PMID 31421023
- [Derived] Gloersen M, Steen Pettersen P, Kvien TK, Haugen IK. Validation of the Intermittent and Constant Osteoarthritis Pain Questionnaire in Patients with Hand Osteoarthritis: Results from the Nor-Hand Study. J Rheumatol. 2019 Jun;46(6):645-651. doi: 10.3899/jrheum.180835. Epub 2019 Mar 15. PMID 30877221
- [Derived] Steen Pettersen P, Neogi T, Magnusson K, Berner Hammer H, Uhlig T, Kvien TK, Haugen IK. Peripheral and Central Sensitization of Pain in Individuals With Hand Osteoarthritis and Associations With Self-Reported Pain Severity. Arthritis Rheumatol. 2019 Jul;71(7):1070-1077. doi: 10.1002/art.40850. Epub 2019 May 14. PMID 30741501
- [Derived] Gloersen M, Mulrooney E, Mathiessen A, Hammer HB, Slatkowsky-Christensen B, Faraj K, Isaksen T, Neogi T, Kvien TK, Magnusson K, Haugen IK. A hospital-based observational cohort study exploring pain and biomarkers in patients with hand osteoarthritis in Norway: The Nor-Hand protocol. BMJ Open. 2017 Sep 24;7(9):e016938. doi: 10.1136/bmjopen-2017-016938. PMID 28947452